CLINICAL TRIAL: NCT02690129
Title: Vaginal Progesterone for Treatment of Threatened Miscarriage; Randomized Clinical Trial
Brief Title: Vaginal Progesterone for Treatment of Threatened Miscarriage
Acronym: VPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omar Mamdouh Shaaban (Other)
Responsible Party: Sponsor-Investigator, Omar Mamdouh Shaaban, Clinical Professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: treatment of miscarraige
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Threatened Miscarriage
Keywords: progesterone; threatened abortion
MeSH Terms: conditions — Abortion, Threatened | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Progesterone Group) (Active Comparator): Complete bed rest as an in/or out- patient, according to patient's preference for first 48-72 hours.
  * Vaginal progesterone treatment as single daily dose of natural micronized progesterone (Prontogest ® 200 mg) at bedtime for 15 days.
  * If needed, a pain killer as Indomethacin 50 mg/ rectally twice daily up to control of uterine colic .
  * Complete abstaining from sexual activity or strenuous effort. Additionally, Rh-ve women with established viable fetuses and continue bleeding will be given a shot of anti-D immunoglobulin 300 ugm/IM ; after 12 weeks' gestation or if undergo surgical evacuation.
  Interventions: Drug: Vaginal Progesteron
- Group II ( Control group) (Placebo Comparator): Will follow the same plan of management without progesterone support.
  Interventions: Drug: Vaginal Progesteron

INTERVENTIONS:
Drug: Vaginal Progesteron
  Other Names: Progesterone

SUMMARY:
The purpose of the study is to assess the efficacy of vaginal micronized progesterone in the treatment of threatened miscarriage. All eligible pregnant women will be randomized to either receive vaginal progesterone or no treatment.Evaluation will be two weeks after intervention, then every 4 weeks up to 28 weeks gestation or termination of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant with gestational age less than 24 weeks
2. Presented by bleeding with or without pain
3. Single viable fetus (confirmed by Ultrasound examination)
4. Accepting to have vaginal medication

Exclusion Criteria:

1. Currently under medication for any chronic diseases (DM, thyroid, liver, renal, cardiac and autoimmune disease).
2. Hypersensitivity to progesterone
3. Any documented congenital fetal anomaly in the current pregnancy
4. Women received hormonal treatment in the current pregnancy
5. Patients conceived via ART

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Miscarriage rate up to 28 weeks of gestation | Completed 28th week

SECONDARY OUTCOMES:
Gestational age at delivery or termination of pregnancy | Number of completed weeks at the time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No